CLINICAL TRIAL: NCT04055025
Title: Physiological Responses to Laparoscopic Sleeve Gastrectomy: Focusing on Ghrelin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Nora Elisabeth Hedbäck, Medical Doctor, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-19010763
Record Dates: First submitted 2019-08-07; First posted 2019-08-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Bariatric Surgery
Keywords: Ghrelin; Sleeve gastrectomy; Laparoscopic sleeve gastrectomy
MeSH Terms: interventions — Ghrelin

STUDY DESIGN:
Masking Description: The study visits will be performed in randomized orders and participants will not now if they will receive ghrelin or saline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleeve gastrectomy operated patients (Other): Six test days in a randomized, patient-blinded, cross-over design
  Interventions: Other: Placebo; Other: Ghrelin

INTERVENTIONS:
Other: Placebo — Four-hour liquid solid meal tests and a subsequent ad libitum meal during saline infusion.
Other: Ghrelin — Four-hour liquid solid meal tests and a subsequent ad libitum meal during acyl-ghrelin infusion.

SUMMARY:
Our hypothesis is that decreased concentration of ghrelin after LSG is important for the decreased appetite and food intake postoperatively. We therefore expect infusion of ghrelin will increase an ad libitum food intake after LSG. We also expect that a decreased postprandial concentration of ghrelin after LSG play a role for increased insulin secretion and decreased postprandial plasma glucose concentrations after surgery.

DETAILED DESCRIPTION:
Laparoscopic Roux-en-Y gastric bypass (LRYGB) and laparoscopic sleeve gastrectomy (LSG) are to bariatric procedure. After both procedures, a changed secretion of hormones from the gastrointestinal tract is believed to affect appetite and glucose metabolism. Studies have shown that after LRYGB, there is a significant increased secretion of GLP-1 and PYY. In contrast, a decreased secretion of ghrelin is a characteristic finding after LSG opposite post-LRYGB, where secretion of ghrelin is reported to be increased, decreased or unchanged. Ghrelin is primarily secreted from the gastric mucosa in the fasting state and decreases in response to food intake. Ghrelin stimulates food intake through appetite-regulating centers in the hypothalamus. Administration of exogenous ghrelin has been reported to stimulate appetite. In addition, ghrelin has recently been suggested also to affect glucose metabolism by inhibition of glucose-stimulated insulin secretion. Therefore the markedly decreased secretion of ghrelin could be of particular important for the decreased appetite and improved glucose tolerance seen after LSG.

ELIGIBILITY:
Inclusion Criteria:

* The Danish national inclusion criteria for bariatric surgery
* Signed written informed consent
* Fasting plasma glucose <6.1 mmol/l

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Hemoglobin <6.5 mM
* Newly emerged serious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Ad libitum | 240 minutes
  Ad libitum food intake (gram) with and without infusion of ghrelin at 3 months after LSG surgery

SECONDARY OUTCOMES:
Ad libitum | 240 minutes
  Ad libitum food intake (gram) with and without ghrelin infusion before surgery.
Ghrelin | 240 minutes
  Plasma concentration profile of ghrelin (AUC) before and after LSG.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Hedbäck, MD, Principal Investigator — Department of Endocrinology, Hvidovre University Hospital, Denmark
Locations (1):
- Department of Endocrinology, Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No